CLINICAL TRIAL: NCT05223920
Title: A Multi-Center, Open Label, Extension Study Evaluating the Safety and Efficacy of Bomedemstat for the Treatment of Patients With Myeloproliferative Neoplasms (MPNs) Enrolled in a Prior Bomedemstat Clinical Study
Brief Title: An Extension Study of Bomedemstat (IMG-7289/MK-3543) in Participants With Myeloproliferative Neoplasms (IMG-7289-CTP-202/MK-3543-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMG-7289-CTP-202; MK-3543-005 (Other: MSD); IMG-7289 (Other: ImagoBio); 2021-002452-37 (EudraCT Number)
Record Dates: First submitted 2021-08-31; First posted 2022-02-04 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Thrombocythemia, Essential; Primary Myelofibrosis
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bomedemstat (Experimental): All participants will receive bomedemstat via oral capsule daily for 169 days with additional treatment continuing in patients deriving clinical benefit.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Capsule (oral)
  Other Names: IMG-7289; MK-3543

SUMMARY:
This is a multi-center, open-label extension study to assess the long-term safety and efficacy of bomedemstat administered orally once daily in participants with a Myeloproliferative Neoplasm (MPN) who participated in a prior bomedemstat study such as, but not limited to, IMG-7289-CTP-102/MK-3543-002 (NCT03136185) and IMG-7289-CTP-201/MK-3543-003 (NCT04254978) (referred to hereafter as 'feeder studies').

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Has completed at least one Treatment Period (TP) in a prior bomedemstat Myeloproliferative Neoplasms (MPN) protocol (such as, but not limited to, IMG-7289-CTP-102/MK-3543-002 (NCT03136185) and IMG-7289-CTP-201/MK-3543-003) (NCT04254978).
* In the estimation of the Investigator, the risk-benefit favors continued dosing with bomedemstat.

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* Ongoing participation in another investigational study (except observational studies).
* A history of non-compliance in a prior bomedemstat study (excluding dose suspensions that were medically warranted).
* Current use of a prohibited medication (e.g., romiplostim).
* Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the patient's safety, ability to give informed consent, or comply with the trial protocol.
* Is pregnant or breastfeeding or plan to become pregnant or breastfeed during the study.
* Women of childbearing potential (WOCBP) and fertile men unwilling to agree to use an approved method of contraception from time of enrollment until 14 days after last bomedemstat dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- United States (5):
  - University of Miami Leonard M. Miller, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UMPC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Gold Coast Hospital and Health Service, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Universittsklinikum Essen, Essen, Germany
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (4):
  - Ospedale di Circolo-a Fondazione Macchi, Varese, VA
  - Azienda Ospedaliera SS. Antonio, Alessandria
  - Azienda Ospedaliero-Universitaria Careggi - S.O.D. Ematologia (CRIMM), Florence
  - Azienda Ospedaliero Universitaria di Bologna, Pavia
- New Zealand (2):
  - Middlemore Clinical Trials, Papatoetoe, Aukland
  - Waitemata District Health Board, Takapuna, Aukland
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and Saint Thomas' NHS Foundation Trus, London

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Myeloproliferative Neoplasms (MPNs) who participated in a prior bomedemstat study such as, but not limited to, IMG-7289-CTP-102/MK-3543-002 (NCT03136185) and IMG-7289-CTP-201/MK-3543-003 (NCT04254978) (referred to hereafter as 'feeder studies') were included in the recruitment.
Pre-assignment Details: Participants were assigned to either the Essential thrombocythemia (ET) arm or Myelofibrosis (MF) arm based on prior diagnosis.
Groups:
- Essential Thrombocythemia (ET): Participants with ET received bomedemstat daily as an oral capsule. The daily dose of bomedemstat was titrated for each participant to a dose that reduced platelets to the target range associated with the participant's underlying MPN.
- Myelofibrosis (MF): Participants with MF received bomedemstat daily as an oral capsule. The daily dose of bomedemstat was titrated for each participant to a dose that reduced platelets to the target range associated with the participant's underlying MPN.
Period: Overall Study
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
Started | 52 | 29
Completed | 0 | 0
Not Completed | 52 | 29
Not completed — Adverse Event | 6 | 3
Not completed — Death | 2 | 0
Not completed — Disease Progression | 1 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Sponsor decision | 11 | 9
Not completed — Transferred to Extension Study MK-3543-017 (NCT06351631) | 29 | 7
Not completed — Subject decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF) | Total
Number analyzed (Participants) | 52 | 29 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (11.01) | 65.3 (9.68) | 65.6 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 14 | 43
  Male | 23 | 15 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 51 | 28 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 35 | 13 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Spleen Volume by Magnetic resonance imaging/computerized tomography (MRI/CT) in mL [Median (Full Range); unit: mL] — Baseline spleen volume was measured for myelofibrosis participants via MRI/CT scan in milliliters (mL). Population: Analysis population contained all MF participants who had baseline measurement.
  mL
    number analyzed (Participants) | 0 | 26 | 26
    (all) |  | 835.21 [98.88 to 3085.92] | 835.21 [98.88 to 3085.92]
Baseline Platelet Counts in thousands per microliter (10^3 cells/μL) [Mean (Standard Deviation); unit: 10^3 cells/μL] — Baseline platelet count measured in 10^3 cells/μL was obtained for both ET and MF participants.
  10^3 cells/μL | 380.4 (207.44) | 190.5 (209.64) | 312.4 (226.29)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience an Adverse Event (AE)
Description: An AE is any undesirable physical, psychological or behavioral effect experienced by a participant during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. This includes any clinically significant abnormalities in vital signs and lab values, untoward signs or symptoms experienced by the participant from the time of first dose with bomedemstat under this protocol until completion of the study. The percentage of participants who experienced an AE is presented.
Time Frame: Up to ~32 months
Population: All participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
Number analyzed (Participants) | 52 | 29
Percentage of Participants | 98.1 | 100.0

2. Primary Outcome: Percentage of Participants Who Discontinue Study Intervention Due to an AE
Description: An AE is any undesirable physical, psychological or behavioral effect experienced by a participant during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. This includes any clinically significant abnormalities in vital signs and lab values, untoward signs or symptoms experienced by the participant from the time of first dose with bomedemstat under this protocol until completion of the study. The percentage of participants who discontinued study intervention due to an AE is presented.
Time Frame: Up to ~32 months
Population: All participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
Number analyzed (Participants) | 52 | 29
Percentage of Participants | 15.4 | 10.3

3. Primary Outcome: Mean Spleen Volume Reduction Based on Spleen Volume Measured by MRI in Participants With MF.
Description: Mean Spleen volume reduction (mL) in participants with MF as measured by central laboratory imaging analysis of MRI (or CT where applicable) approximately every 48 weeks. Per protocol only participants with MF were analyzed for this outcome measure. The change in spleen volume from baseline is presented.
Time Frame: Baseline and Days 169, 339, 509, 679, 849 and 924
Population: The modified intent to treat (mITT) population included all participants who were enrolled in the study, received at least 1 dose of study intervention, and who had a nonmissing baseline and at least 1 nonmissing postbaseline efficacy assessment. Participants were analyzed according to treatment received in the study. Per protocol only participants with MF were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
Number analyzed (Participants) | 0 | 29
mL
  Day 169: number analyzed (Participants) | 0 | 2
  Day 169 |  | -101.570 (92.6876)
  Day 339: number analyzed (Participants) | 0 | 16
  Day 339 |  | -67.645 (249.0079)
  Day 509: number analyzed (Participants) | 0 | 3
  Day 509 |  | -5.920 (143.1692)
  Day 679: number analyzed (Participants) | 0 | 15
  Day 679 |  | -61.000 (396.2520)
  Day 849: number analyzed (Participants) | 0 | 1
  Day 849 |  | -38.840 (NA) — Standard deviation is not estimable due to only 1 participant in the group.
  Day 924: number analyzed (Participants) | 0 | 2
  Day 924 |  | 80.575 (10.3308)

4. Primary Outcome: Percentage of Participants With ET Who Achieve a Reduction of Platelet Counts to <= 400 K/uL (400 x 10^9/L) in the Absence of New Thromboembolic Events
Description: Blood samples were taken at designated time points to determine platelet count. Percentage of participants with ET who achieve a reduction of platelet counts to <= 400 K/uL (400 x 10^9/L) in the absence of new thromboembolic events is presented.
Time Frame: Baseline and Days 29, 57, 85, 113, 141, 169, 198, 226, 254, 282, 310, 338, 367, 395, 423, 451, 479, 507, 536, 564, 592, 620, and 648
Population: The modified intent to treat (mITT) population included all participants who were enrolled in the study, received at least 1 dose of study intervention, and who had a nonmissing baseline and at least 1 nonmissing postbaseline efficacy assessment. Per protocol only participants with ET were analyzed for this outcome measure. Participants were analyzed according to treatment received in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
Number analyzed (Participants) | 52 | 0
Percentage of participants
  Day 29: number analyzed (Participants) | 48 | 0
  Day 29 | 77.1 [62.7 to 88.0] |
  Day 57: number analyzed (Participants) | 48 | 0
  Day 57 | 72.9 [58.2 to 84.7] |
  Day 85: number analyzed (Participants) | 50 | 0
  Day 85 | 72.0 [57.5 to 83.8] |
  Day 113: number analyzed (Participants) | 51 | 0
  Day 113 | 78.4 [64.7 to 88.7] |
  Day 141: number analyzed (Participants) | 49 | 0
  Day 141 | 91.8 [80.4 to 97.7] |
  Day 169: number analyzed (Participants) | 47 | 0
  Day 169 | 89.4 [76.9 to 96.5] |
  Day 198: number analyzed (Participants) | 45 | 0
  Day 198 | 86.7 [73.2 to 94.9] |
  Day 226: number analyzed (Participants) | 44 | 0
  Day 226 | 81.8 [67.3 to 91.8] |
  Day 254: number analyzed (Participants) | 44 | 0
  Day 254 | 79.5 [64.7 to 90.2] |
  Day 282: number analyzed (Participants) | 44 | 0
  Day 282 | 75.0 [59.7 to 86.8] |
  Day 310: number analyzed (Participants) | 43 | 0
  Day 310 | 81.4 [66.6 to 91.6] |
  Day 338: number analyzed (Participants) | 43 | 0
  Day 338 | 83.7 [69.3 to 93.2] |
  Day 367: number analyzed (Participants) | 42 | 0
  Day 367 | 76.2 [60.5 to 87.9] |
  Day 395: number analyzed (Participants) | 41 | 0
  Day 395 | 78.0 [62.4 to 89.4] |
  Day 423: number analyzed (Participants) | 40 | 0
  Day 423 | 80.0 [64.4 to 90.9] |
  Day 451: number analyzed (Participants) | 39 | 0
  Day 451 | 82.1 [66.5 to 92.5] |
  Day 479: number analyzed (Participants) | 37 | 0
  Day 479 | 75.7 [58.8 to 88.2] |
  Day 507: number analyzed (Participants) | 26 | 0
  Day 507 | 96.2 [80.4 to 99.9] |
  Day 536: number analyzed (Participants) | 19 | 0
  Day 536 | 94.7 [74.0 to 99.9] |
  Day 564: number analyzed (Participants) | 15 | 0
  Day 564 | 86.7 [59.5 to 98.3] |
  Day 592: number analyzed (Participants) | 11 | 0
  Day 592 | 72.7 [39.0 to 94.0] |
  Day 620: number analyzed (Participants) | 7 | 0
  Day 620 | 85.7 [42.1 to 99.6] |
  Day 648: number analyzed (Participants) | 6 | 0
  Day 648 | 83.3 [35.9 to 99.6] |

ADVERSE EVENTS:
Time Frame: Death and adverse events up to ~32 months
Description: All-cause mortality was reported on all allocated participants. Serious and non-serious adverse events (AEs) were reported on all participants who received ≥1 dose of study treatment.
Arm/Group | Essential Thrombocythemia (ET) | Myelofibrosis (MF)
All-Cause Mortality (participants affected / at risk) | 2/52 | 0/29
Serious Adverse Events (participants affected / at risk) | 19/52 | 12/29
Other Adverse Events (participants affected / at risk) | 45/52 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essential Thrombocythemia (ET) (N=52) | Myelofibrosis (MF) (N=29)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Wellens' syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essential Thrombocythemia (ET) (N=52) | Myelofibrosis (MF) (N=29)
Anaemia (Blood and lymphatic system disorders) | 10 (11) | 7 (16)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (13) | 12 (27)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (9) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (5) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 7 (8)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 3 (3) | 7 (14)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (10)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (5)
Fatigue (General disorders) | 7 (8) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 3 (4) | 2 (3)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 11 (15)
Cellulitis (Infections and infestations) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 4 (5)
Urinary tract infection (Infections and infestations) | 7 (8) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 6 (13)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 3 (8) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 4 (4)
Urinary occult blood (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (24) | 14 (21)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 7 (7) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 3 (5) | 3 (3)
Hypertension (Vascular disorders) | 4 (7) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT05223920/Prot_SAP_000.pdf